CLINICAL TRIAL: NCT07401017
Title: The Effects of Rosuvastatin on Physiological Adaptation and Safety During Regular Long-Distance Running Training: A Randomized Controlled Trial
Brief Title: The Effects of Rosuvastatin on Running Training Adaptation and Safety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: N2025102501
Record Dates: First submitted 2025-12-01; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Dyslipidemia; Long-Distance Running; Endurance Training; Statin-Associated Muscle Symptoms
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin group (Experimental)
  Interventions: Drug: Rosuvastatin
- Control group (No Intervention)

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 10 mg tablet taken orally once daily at bedtime for 3 months.
  Arms: Rosuvastatin group

SUMMARY:
Statins lower low-density lipoprotein cholesterol (LDL-C) and help prevent atherosclerotic cardiovascular disease, but some users develop statin-associated muscle symptoms (SAMS) such as soreness, stiffness, weakness, or elevated creatine kinase (CK). These symptoms may be more noticeable during exercise. Regular long-distance running improves cardiopulmonary fitness-VO₂max, aerobic threshold (AT), and respiratory compensation point (RCP)-mainly through mitochondrial and metabolic adaptations. Prior studies suggest that lipophilic statins like simvastatin may blunt these adaptations, while hydrophilic statins such as rosuvastatin may have a smaller impact. However, prospective data in habitual endurance runners are limited.

This randomized controlled trial will examine how rosuvastatin affects cardiopulmonary fitness improvements and muscle tolerance in individuals who run at least three times per week and meet clinical criteria for statin therapy. After informed consent and baseline cardiopulmonary exercise testing (CPET), participants will be randomized to rosuvastatin 10 mg daily or no statin therapy for three months. Both groups will maintain their usual training routines, and training load will be recorded using heart-rate-based TRIMP. CPET will be repeated monthly to assess changes in VO₂max, AT, and RCP, and muscle enzymes and SAMS will be evaluated at each visit.

The study aims to clarify whether rosuvastatin influences endurance-related physiological adaptations or increases muscle symptoms in regular long-distance runners.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Meets clinical criteria for statin therapy, including at least one of the following:
* Family history of hyperlipidemia.
* LDL-C ≥ 160 mg/dL.
* 10-year Atherosclerotic Cardiovascular Disease (ASCVD) risk ≥ 7.5%
* Diabetes mellitus with LDL-C ≥ 70 mg/dL.
* Determined by a clinician to require lipid-lowering therapy.
* Currently using or eligible to initiate rosuvastatin therapy.
* Performs long-distance running at least 3 times per week and is willing to maintain regular training for 3 months.
* Able and willing to undergo cardiopulmonary exercise testing (CPET) and to record training data using a sports watch (for TRIMP calculation).
* No known drug allergies and provides written informed consent after study explanation.

Exclusion Criteria:

* Known allergy or intolerance to statins or rosuvastatin.
* History of severe statin-related adverse events, including rhabdomyolysis or marked creatine kinase (CK) elevation.
* Liver dysfunction with AST or ALT > 3× upper limit of normal.
* Moderate to severe renal impairment (eGFR < 30 mL/min/1.73 m²).
* Current lower-limb pain, tendon injury, or other conditions that prevent running training.
* Not suitable for maximal cardiopulmonary exercise testing (CPET), such as unstable angina, uncontrolled hypertension, or recent cardiovascular events.
* Pregnant or breastfeeding.
* Inability to comply with study procedures, including use of a sports watch, regular follow-up visits, or maintaining running training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
VO₂max (mL/kg/min) | Baseline (Month 0), Month 1, Month 2, Month 3
  Maximum oxygen consumption obtained from cardiopulmonary exercise testing (CPET). Used to assess changes in cardiopulmonary fitness over the 3-month intervention period.
Aerobic Threshold (AT) | Baseline, Month 1, Month 2, Month 3
  Aerobic threshold determined by standardized CPET. Represents the transition from aerobic to anaerobic metabolism during exercise.
Respiratory Compensation Point (RCP) | Baseline, Month 1, Month 2, Month 3
  RCP measured via CPET, representing the ventilatory response to metabolic acidosis. Used to evaluate endurance training adaptation.

SECONDARY OUTCOMES:
Calculated Training Load Score (using TRIMP method) | Through the end of the 3-month intervention period
  Training load is reported as a single Training Impulse (TRIMP) score. It is calculated by multiplying exercise duration (minutes) by a heart-rate-based intensity factor (e.g., fractional heart rate reserve). This integrates two metrics into one unified numerical value.
  The formula is: TRIMP = Duration (min) x [ΔHR ratio] x y
  Where:
  ΔHR ratio = (HR_ex - HR_rest) / (HR_max - HR_rest) y = A weighting factor derived from an exponential function to account for the disproportionate increase in physiological strain at higher exercise intensities (using gender-specific constants: 0.64e^(1.92x) for males and 0.86e^(1.67x) for females).
Number of Participants with Statin-Associated Muscle Symptoms (SAMS) | Month 1, Month 2, and Month 3
  Number of participants reporting any muscle soreness, weakness, or stiffness as assessed by the SAMS questionnaire.
Change from Baseline in Body Weight (kg) | Baseline, Month 1, Month 2, Month 3
  Body weight measured in kilograms (kg) to evaluate changes during the training and intervention period.
Change from Baseline in Body Mass Index (kg/m^2) | Baseline, Month 1, Month 2, Month 3
  Body Mass Index (BMI) calculated as weight in kilograms divided by height in meters squared (kg/m^2).

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsuan Cheng, MD, MS, Study Chair — Taipei Medical University
Locations (1):
- Taipei medical university, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sigrist C, Murner-Lavanchy I, Peschel SKV, Schmidt SJ, Kaess M, Koenig J. Early life maltreatment and resting-state heart rate variability: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2021 Jan;120:307-334. doi: 10.1016/j.neubiorev.2020.10.026. Epub 2020 Nov 7. PMID 33171141
- [Background] Glei M, Schlormann W. Analysis of DNA damage and repair by comet fluorescence in situ hybridization (Comet-FISH). Methods Mol Biol. 2014;1094:39-48. doi: 10.1007/978-1-62703-706-8_4. PMID 24162978
- [Background] Yamada Y, Hoyano M, Akashi R, Oto K, Kanemitsu Y. Impact of Chemical Doping on Optical Responses in Bismuth-Doped CH3NH3PbBr3 Single Crystals: Carrier Lifetime and Photon Recycling. J Phys Chem Lett. 2017 Dec 7;8(23):5798-5803. doi: 10.1021/acs.jpclett.7b02508. Epub 2017 Nov 15. PMID 29130309
- [Background] Najmeddin F, Khalili H. Comment on: Guidelines for the diagnosis and antibiotic treatment of endocarditis in adults: a report of the Working Party of the British Society for Antimicrobial Chemotherapy. J Antimicrob Chemother. 2012 Dec;67(12):3016-7; author reply 3017. doi: 10.1093/jac/dks290. Epub 2012 Jul 24. No abstract available. PMID 22833643
- [Background] Tabit CE, Shenouda SM, Holbrook M, Fetterman JL, Kiani S, Frame AA, Kluge MA, Held A, Dohadwala MM, Gokce N, Farb MG, Rosenzweig J, Ruderman N, Vita JA, Hamburg NM. Protein kinase C-beta contributes to impaired endothelial insulin signaling in humans with diabetes mellitus. Circulation. 2013 Jan 1;127(1):86-95. doi: 10.1161/CIRCULATIONAHA.112.127514. Epub 2012 Nov 30. PMID 23204109
- [Background] Park JS, Park D. Effect of Polydeoxyribonucleotide Injection in a Patient With Carpal Tunnel Syndrome. Am J Phys Med Rehabil. 2018 Oct;97(10):e93-e95. doi: 10.1097/PHM.0000000000000901. PMID 29373371
- [Background] Hartiala O, Magnussen CG, Kajander S, Knuuti J, Ukkonen H, Saraste A, Rinta-Kiikka I, Kainulainen S, Kahonen M, Hutri-Kahonen N, Laitinen T, Lehtimaki T, Viikari JS, Hartiala J, Juonala M, Raitakari OT. Adolescence risk factors are predictive of coronary artery calcification at middle age: the cardiovascular risk in young Finns study. J Am Coll Cardiol. 2012 Oct 9;60(15):1364-70. doi: 10.1016/j.jacc.2012.05.045. Epub 2012 Sep 12. PMID 22981553
- [Background] Mikus CR, Boyle LJ, Borengasser SJ, Oberlin DJ, Naples SP, Fletcher J, Meers GM, Ruebel M, Laughlin MH, Dellsperger KC, Fadel PJ, Thyfault JP. Simvastatin impairs exercise training adaptations. J Am Coll Cardiol. 2013 Aug 20;62(8):709-14. doi: 10.1016/j.jacc.2013.02.074. Epub 2013 Apr 10. PMID 23583255